CLINICAL TRIAL: NCT05846854
Title: Novel Protocol to Decrease Peri-procedural and Intra-operative Hemorrhage in Children With Alagille Syndrome
Brief Title: Decreasing Hemorrhage Risk in Children With Alagille Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Stanford University (Other)
Collaborators: Alagille Syndrome Alliance (Unknown)
Responsible Party: Principal Investigator, Noelle Hanako, Associate Professor, Division of Pediatric Gastroenterology, Hepatology and Nutrition, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 66477
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Alagille Syndrome; Pulmonary Artery Stenoses; Acquired Von Willebrand Disease
MeSH Terms: conditions — Alagille Syndrome; Stenosis, Pulmonary Artery | interventions — Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alagille syndrome (Experimental): Patients with complex cardiac conditions requiring cardiothoracic surgery who also have a history of Alagille syndrome.
  Interventions: Other: Assessment for bleeding disorder with tailored post-operative care
- No history of Alagille syndrome (Experimental): Patients with complex cardiac conditions requiring cardiothoracic surgery who do not have a diagnosis of Alagille syndrome.
  Interventions: Other: Assessment for bleeding disorder with tailored post-operative care

INTERVENTIONS:
Other: Assessment for bleeding disorder with tailored post-operative care — Intervention will be expanded lab work-up for hematologic conditions, consultation by Hematology and tailored intra-operative and post-operative plan with aim to mitigate bleeding and hemorrhage risk, balancing thrombotic risk with this intervention.

SUMMARY:
The goal of this interventional study is to test a hemostasis screening protocol and cardiac peri-procedural and post-operative hemostasis pathway to improving bleeding complications and improve patient survival for children with Alagille syndrome and complex cardiac conditions. The main questions it aims to answer are:

* Are children with Alagille syndrome with cardiac anomalies more likely to have acquired von Willebrand syndrome (a condition that causes increased bleeding)
* Does implementation of a novel screening protocol to detect pre-operative bleeding conditions decrease intra-operative and/or post-operative bleeding complications and mortality risk?
* Does implementation of a novel screening protocol to detect and treat bleeding conditions cause thrombotic complications?

Participants will undergo additional hematology and bleeding disorder screening prior to cardiac surgery. They will additionally undergo a detailed family screening for a history of bleeding by a genetic counselor.

Researchers will compare these findings with children who have similar complex cardiac conditions requiring surgery, but who do not have Alagille syndrome to see if bleeding conditions and complications are more or less common in children with Alagille syndrome.

DETAILED DESCRIPTION:
This study aims to develop and implement a pre-operative screening protocol prior to major procedures or surgeries for children with Alagille syndrome, including cardiac catheterization and cardiothoracic surgery (pulmonary artery reconstruction).

Secondary Objectives

1. Develop and implement an intra-operative protocol for children with Alagille syndrome and acquired von willebrand syndrome.
2. Compare cardiac intra- and up to 48 hour post-operative bleeding complications, post-operative thrombotic complications within 30 days of surgery, and mortality for (a) children with Alagille syndrome with and without acquired von willebrand syndrome, and (b) children without Alagille syndrome.

This is a single-site study with the goal to enroll 40 patients over the course of the study period. All patients that are referred for Pulmonary Artery Reconstruction will be screened for eligibility. All patients will undergo standard of care pre-operative hematologic screening to evaluate for bleeding disorders (specifically platelet aggregation disorders and acquired von Willebrand Factor deficiency).

The study includes a pre-screening period of up to 4 weeks followed by a 12-months follow-up period as part of the standard of care following pulmonary artery reconstruction surgery for children with Alagille syndrome and a research related protocol for children without Alagille syndrome.

Patients would have blood drawn one time at least 2 weeks in advance of their cardiothoracic surgery. This is the screening protocol to understand if they have a bleeding disorder that would change their management in the operating room and after their surgery. For patients that are found to have a bleeding disorder requiring treatment, they would need post-operatively a blood test daily for up to 7 days total and another blood test weekly for 2 weeks and then once prior to discharge.

ELIGIBILITY:
Inclusion Criteria:

* 0-17 years old
* with complex cardiac condition requiring pulmonary artery reconstruction (branch pulmonary artery stenosis, MAPCAs or Tetralogy of Fallot without MAPCAs)

Exclusion Criteria:

* history of known bleeding disorder
* aged 18 years or older

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Blood product volume | Intra-operatively through 24 hours post-operatively
Chest tube output blood volume | Intra-operatively through 24 hours post-operatively
Number of participants with pulmonary hemorrhage | Intra-operatively through 24 hours post-operatively

SECONDARY OUTCOMES:
Incidence of thromboembolism events in patients with hematologic condition | Intra-operatively through 30 days post-operatively
  This outcome is to evaluate thrombosis risk for patients identified to have a hematologic condition who receive medication intra-operatively and post-operatively to decrease their risk of bleeding. Occurrence of thromboembolism (including blood vessel, intracardiac, stroke, mediastinal thrombosis events) will be assessed based on imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Noelle Ebel, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No